CLINICAL TRIAL: NCT03291795
Title: Prehabilitation Exercise Plus Perioperative Optimization of Senior Health
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: feasibility challenges
Sponsor: Duke University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00076925; P30AG028716 (NIH)
Record Dates: First submitted 2017-09-13; First posted 2017-09-25 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-06

CONDITIONS: Cognitive Decline; Age-Related Memory Disorders; Postoperative Complications; Age-Related Atrophy; Postoperative Cognitive Dysfunction
MeSH Terms: conditions — Cognitive Dysfunction; Memory Disorders; Postoperative Complications; Postoperative Cognitive Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise Intervention (Experimental)
  Interventions: Other: Exercise Intervention

INTERVENTIONS:
Other: Exercise Intervention — Study patients will undergo a program of prehabilitation exercise for 6 days per week prescribed for them by an exercise physiologist, for up to 4 weeks prior to surgery.

SUMMARY:
The purpose of this study is the examine the feasibility of and estimate the efficacy of a preoperative exercise (i.e. prehabilitation) program in 40 up to sedentary older adults (i.e. age 60 and over) undergoing abdominal, urologic or gynecologic surgery under the Enhanced Recovery After Surgery (ERAS) protocol at Duke, using a variety of techniques to measure the possible effect of this intervention. Study patients will undergo a program of prehabilitation exercise for 6 days per week prescribed for them by an exercise physiologist, for up to 4 weeks prior to surgery. Study participants will undergo four types of assessments: Functional/Cognitive testing; Blood/cerebrospinal fluid (CSF) samples and Muscle biopsies; Brain Imaging; and Brain Activity Recording. Clinical Outcomes will also be obtained from the Duke electronic medical record system. The risks of the exercise intervention are generally mild, since moderate exercise in this patient population generally results in improved health outcomes. Data from these patients will be analyzed in comparison to propensity matched patients from the Duke Markers of Alzheimer's Disease and neurocognitive Outcomes after Perioperative Care (MADCO-PC) study who did not undergo this prehabilitation exercise intervention. Taken together, the results of this study will allow the investigators to estimate the possible effect of prehabilitation exercise on multiple domains of postoperative recovery (cognition, brain connectivity, biomarkers, brain activity, etc) and will provide important preliminary data.

DETAILED DESCRIPTION:
The purpose of this study is the examine the feasibility of and estimate the efficacy of a preoperative exercise (i.e. prehabilitation) program in 40 up to sedentary older adults (i.e. age 60 and over) undergoing abdominal, urologic or gynecologic surgery under the Enhanced Recovery After Surgery (ERAS) protocol at Duke, using a variety of techniques to measure the possible effect of this intervention. Study patients will undergo a program of prehabilitation exercise for 6 days per week prescribed for them by an exercise physiologist, for up to 4 weeks prior to surgery. Study participants will undergo four types of assessments: Functional/Cognitive testing; Blood/CSF samples and Muscle biopsies; Brain Imaging; and Brain Activity Recording. Clinical Outcomes will also be obtained from the Duke electronic medical record system. The risks of the exercise intervention are generally mild, since moderate exercise in this patient population generally results in improved health outcomes. Data from these patients will be analyzed in comparison to propensity matched patients from the Duke Markers of Alzheimer's Disease and neurocognitive Outcomes after Perioperative Care (MADCO-PC) study who did not undergo this prehabilitation exercise intervention. Taken together, the results of this study will allow the investigators to estimate the possible effect of prehabilitation exercise on multiple domains of postoperative recovery (cognition, brain connectivity, biomarkers, brain activity, etc) and will provide important preliminary data and will help design future more definitive studies to test these hypotheses.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 and above
* Able to speak English.
* seen, scheduled to be seen, or eligible to be seen in Preoperative Optimization of Senior Health (POSH) clinic prior to surgery
* scheduled for general, gynecologic or urologic surgery under the Enhanced Recovery After Surgery (ERAS) protocol, or eligible for ERAS protocol
* Lives within a ~1 hr drive of Duke
* Sedentary (not currently following physical activity guidelines)
* Ambulatory (assistive devices ok)
* Able to give informed consent
* Willing to perform prescribed exercises

Exclusion Criteria:

* Inmate of a correctional facility (i.e. prisoners).
* Documented or suspected family or personal history of malignant hyperthermia.
* Allergy or other contraindication to receiving isoflurane
* Receiving systemic chemotherapy after the first cognitive testing session and before the 6 wk follow up cognitive testing sessions.
* Major head trauma that occurs after the first cognitive testing session and before the 6 wk follow up cognitive testing sessions.
* Anginal symptoms, known coronary artery disease (CAD), or high cardiovascular risk per American College of Cardiology (ACC)/ American Heart Association (AHA) guidelines
* Taking anticoagulants that would preclude lumbar puncture per the American Society of Regional Anesthesia guidelines.
* Diagnosed history of dementia.
* Inability to ambulate independently.
* Otherwise not appropriate for study participation in the judgement of the Principal Investigator, such as (but not limited to) because the patient does not have the cardiopulmonary capacity to complete the exercise regimen.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-08-20 (Actual); Primary Completion 2018-01-08 (Actual); Study Completion 2018-01-08 (Actual)

PRIMARY OUTCOMES:
Feasibility of Preoperative exercise program | approximately 18 months
  The number of patients contacted versus the number of patients enrolled will be tracked to determine recruitment feasibility. Reasons for refusal will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Miles Berger, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided